CLINICAL TRIAL: NCT05309980
Title: Outcomes in CArdiogenic SHock Patients Treated by MEchanical Circulatory suppoRt devicE : Impact of Shock Team
Acronym: CASHMERE
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Principal Investigator, Alexandre OUATTARA, MD, PhD, University Hospital, Bordeaux
Other Study IDs: CHUBX2020RE0273
Record Dates: First submitted 2021-12-08; First posted 2022-04-04 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2022-03

CONDITIONS: Cardiogenic Shock; Short Term Mechanical Circulatory Support; Shock Team
Keywords: Extra Corporeal Membrane Oxygenation; Cardiogenic Shock; Impella; Shock Team; Long Term Mechanical Circulatory Support
MeSH Terms: conditions — Shock, Cardiogenic | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Without Shock Team: Before January 2013, patients with refractory cardiogenic shock were implanted with short term mechanical circulatory device without involvment of a dedicated shock team
  Interventions: Other: standard of care
- With Shock Team: After April 2013, patients with refractory cardiogenic shock were implanted with short term mechanical circulatory device following a collegial meeting of a shock team (cardiac surgeon, cardiologist, intensivist) using a common algorythm.
  Interventions: Other: standard of care

INTERVENTIONS:
Other: standard of care — retrospective study : standard of care

SUMMARY:
In this before-after monocenter study, the authors teste the hypothesis that the implementation of a dedicated shock team could improve the outcome of patients with refractory cardiogenic shock assisted by mechanical circulatory support.

DETAILED DESCRIPTION:
Short Term Mechanical Circulatory Support (STMCS) are the last resort therapeutics when refractory cardiogenic shock occurs. Growing technical possibilities like impella make the right choice at the right time challenging. At Bordeaux University Hospital, we have gathered the main protagonists which are the surgeon, the interventional cardiologist,and the intensivist as a shock team in January 2013. From that time, diagnosis of refractory cardiogenic shock triggers a multidisciplinary meeting driven by a common algorithm. The objective of this study is to perform a before-after comparison between decision of STMCS for refractory cardiogenic shock without shock team from january 2007 to january 2013 and after implementation of the shock team from April 2013 to April 2019.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cardiogenic shock
* >1 sign of refractory cardiogenic shock : Dobutamine >10µg/kg/mn, epinephrine>0.25µg/kg/mn or Milrinone > 0.5µg/kg/mn ; ScvO2<55% ; pO2/FiO2<100
* No major counter indication to short term mechanical circulatory support : SOFA score > 15, prolonged cardiac arrest, severe chronic disease, direct LVAD implantation or heart transplantation, counter indication for systemic anticoagulation

Exclusion Criteria:

* Age < 18years
* Post cardiotomy cardiogenic shock
* Implantation of Impella 2.5 alone
* Implantation of Intra Aortic Balloon Pump alone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with refractory cardiogenic shock treated with short term mechanical circulatory support between January 2007 to April 2019. A two months wash out period following shock team initiation (February and March 2013) has been set.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Vital status | One year after short term mechanical circulatory support initiation
  Proportion of patients alive

SECONDARY OUTCOMES:
Vital status | 30 days after short term mechanical circulatory support initiation
  proportion of patients alive
Vital status | 3 months after short term mechanical circulatory support initiation
  proportion of patients alive
Vital status | 6 months after short term mechanical circulatory support initiation
  proportion of patients alive
Lenght of stay | up to Intensive Care Unit discharge, an average of 15 days
  Intensive Care Unit length of stay
Lenght of stay | up to one year
  Hospital length of stay
Long term mechanical circulatory support | up to intensive care unit discharge, an average of 15 days
  proportion of patients bridged to long term mechanical circulatory support
Heart transplantation | up to intensive care unit discharge, an average of 15 days
  proportion of patients bridged to heart transplantation
Weaning from short term mechanical circulatory support | up to seven days from weaning attempt
  proportion of patients sucessfully weaned from short term mechanical circulatory support
New renal replacement therapy | up to intensive care unit discharge, an average of 15 days
  proportion of patients needing renal replacement therapy
Limb ischaemia | through short term mechanical circulatory support weaning, an average of 6 days
  proportion of patients with limb ischaemia
Stroke | through short term mechanical circulatory support weaning, an average of 6 days
  proportion of patients with stroke
Short term mechanical circulatory support duration | through short term mechanical circulatory support weaning, an average of 6 days
  Short term mechanical circulatory support duration
Severe haemorrage | through short term mechanical circulatory support weaning, an average of 6 days
  proportion of patients with severe haemorrage (massive haemorrhage according to SFAR or use of Novoseven or rescue surgery for bleeding)
Extra Corporeal Membrane Oxygenation circuit clotting | through short term mechanical circulatory support weaning, an average of 6 days
  proportion of patients in which Extra Corporeal Membrane Oxygenation circuit clotting occured
Sepsis | up to intensive care unit discharge, an average of 15 days
  proportion of patients in which sepsis occured
Vital status | One year after short term mechanical circulatory support initiation
  proportion of patients alive when bridged to long term mechanical circulatory device or when transplanted
Vital status | 30 days after short term mechanical circulatory support initiation
  proportion of patients alive when bridged to long term mechanical circulatory device or when transplanted
Vital status | 3 months after short term mechanical circulatory support initiation
  proportion of patients alive when bridged to long term mechanical circulatory device or when transplanted
Vital status | 6 months after short term mechanical circulatory support initiation
  proportion of patients alive when bridged to long term mechanical circulatory device or when transplanted

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Ouattara, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Bordeaux University Hospital, Pessac, France